CLINICAL TRIAL: NCT00557037
Title: A Phase II Trial of Phenoxodiol in Patients With Castrate and Non-Castrate Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MEI Pharma, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yale 0703002467
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Prostate Cancer
Keywords: Castrate and Non-Castrate Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — phenoxodiol

ARMS (2):
- A (Experimental): Patients with chemotherapy naïve androgen independent disease
  Interventions: Drug: Phenoxodiol
- B (Experimental): Patients with rising PSA after radical prostatectomy or radiotherapy that are androgen dependent
  Interventions: Drug: Phenoxodiol

INTERVENTIONS:
Drug: Phenoxodiol — Oral capsule, 400 mg every 8 hours daily, for 12 weeks - assement to a maximum of 12 months

SUMMARY:
Two groups of patients with prostate cancer will be enrolled:

Group A: patients whose cancer has worsened or spread after being on hormonal therapy and has not had any chemotherapy.

Group B: patients who have a rising PSA after surgery or radiotherapy for the prostate and do not have any spread to the bones or other organs.

Patients will receive Phenoxodiol (PXD) 400 mg every 8 hours daily for 28 consecutive days (1 cycle). Treatment outcome will be evaluated after three cycles (12 weeks) of PXD treatment (immediately prior to cycle 4). Patients with progression of disease will be taken off study. Responding and stable disease patients will remain on study for a total of 12 cycles(approximately 12 months).

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed adenocarcinoma of the prostate
* Patients with castrate and non-castrate levels of testosterone are eligible as defined below.
* Patients with castrate level of testosterone (Group A- androgen independent disease) need to meet the following criteria:
* Progressive disease based on any one of the following

  a) a rise in PSA, b) transaxial imaging, or c) radionuclide bone scan. Patients whose sole manifestation of progression is an increase in disease related symptoms are not eligible.
  1. PSA - a minimum of 3 consecutive rising levels, with an interval of > 1 week between each determination. The last determination must have a minimal value of > 4 ng/ml and be determined within two weeks prior to registration.
  2. Measurable Disease: Patient showing new or progressive soft tissue masses on CT or MRI scans are eligible.
  3. Radionuclide bone scan: New metastatic lesions.
* Serum testosterone < 50 ng/ml, determined within two weeks prior to starting treatment
* Maintaining castrate status: Patients who have not undergone surgical orchiectomy should continue on medical therapies [i.e. gonadotropin releasing hormone analogs (GnRH analogs) to maintain castrate levels of serum testosterone. Patients who are receiving an anti-androgen as part of their first-line hormonal therapy must have shown progression of disease off of the anti-androgen prior to enrollment. Patients must discontinue Megestrol Acetate (MEGACE) and show progression of disease off of this medication.
* No prior chemotherapy except for adjuvant or neo-adjuvant therapy given > than 3 years prior to enrollment
* No more than one prior course of palliative radiotherapy. No prior radioisotope therapy with Strontium-89 or Samarium.
* Patients with non-castrate levels of testosterone (Group B- androgen dependent disease) need to meet the following criteria:
* A rising PSA after radical prostatectomy, radiotherapy or radiation implants with no evidence of metastatic disease on bone, CT scan or MRI scan.
* PSA doubling time less than 12 months
* Testosterone level > 50 ng/ml
* Age > 18 years of age.
* Karnofsky Performance Status > 70%
* Four weeks since major surgery.
* Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment.
* Required Initial Laboratory Data:

  * WBC > 3,000/µl
  * ANC > 1,500/µl
  * Hemoglobin > 9 g/dl
  * Platelet count > 100,000/µl
  * Creatinine < 1.5 x upper limits of normal
  * Bilirubin within 2 x normal limits
  * SGOT (AST) < 2.5 x upper limits of normal
  * SGPT (AST) < 2.5 x upper limits of normal
  * PSA > 4.0 ng/ml (if no measurable disease for Group B) > 4.0 ng/ml for Group A
  * PT within normal limits(*)
  * PTT within normal limits(*)

(*)unless patients are already anti-coagulated for other reasons (i.e. atrial fibrillation, etc.)

* Agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation and for additional 1 months after finishing Phenoxodiol.
* Able to swallow and retain oral medication
* Life expectancy >3 months

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients may continue on a daily Multi-Vitamin and Calcium supplements but all other herbal, alternative and food supplements (i.e. PC-Spes, Saw Palmetto, St John Wort, etc.) must be discontinued before registration.
* Bisphosphonate therapy for bone metastases is allowed; however, treatment must be initiated prior to the first dose of PXD. Prophylactic use of bisphosphonates in patients without bone disease, except for the treatment of osteoporosis, and initiation of bisphosphonates during study treatment is not permitted.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris or recent myocardial infarction (within the last 6 months) are excluded.
* Patients with prior history of hemorrhagic or thrombotic cerebral vascular accident, deep venous thrombosis or pulmonary embolism within the past 6 months are excluded.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not to be registered. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered (by their physician) to be at less than 30% risk for relapse.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with Phenoxodiol. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that have a 50% post-therapy PSA decline at 12 weeks in patients with: a)Chemotherapy naïve androgen independent disease (Group A) b)Rising PSA after radical prostatectomy or radiotherapy that are androgen dependent (Group B) | 12 weeks

SECONDARY OUTCOMES:
To determine the proportion of patients treated with Phenoxodiol that has measurable disease regression at 12 weeks in patients with chemotherapy naïve androgen independent disease. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kelly, MD, Principal Investigator — Yale New Haven Hospital
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut